CLINICAL TRIAL: NCT03249844
Title: High Dose Steroids in Children With Stroke and Unilateral Focal Arteriopathy: Paediatric Arteriopathy Steroid Aspirin (PASTA) Project. A Multicentre Randomized Trial.
Brief Title: Paediatric Arteriopathy Steroid Aspirin Project
Acronym: PASTA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: discontinuation of the trial
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1608184; 2017-002247-15 (EudraCT Number)
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Arterial Ischemic Stroke
Keywords: arterial ischemic stroke; children; steroids; aspirin; Methylprednisolone; Prednisolone
MeSH Terms: conditions — Ischemic Stroke | interventions — Methylprednisolone; Prednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor don't know patient treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Children will be treated by methylprednisolone + prednisolone and standard of care
  Interventions: Drug: Methylprednisolone + prednisolone
- control group (No Intervention): Children will be treated by standard of care alone

INTERVENTIONS:
Drug: Methylprednisolone + prednisolone — The experimental intervention consists of 5 consecutive days Methylprednisolone at a daily single intravenous dose of 20 mg/kg body-weight (max 1 g/day) followed by a 4-week course of tapering Prednisolone given at a daily single oral dose in the morning:
  * week 1 and 2, oral Prednisolone 1 mg/kg/day (max 40 mg/day), ,
  * week 3 and 4, oral Prednisolone 0,5 mg/kg/day (max 20 mg/day),
  Arms: experimental group

SUMMARY:
Arterial ischemic stroke (AIS) is a devastating condition, affecting 1.6-5/100,000 children/year. Although their outcome is different, children with stroke do not recover better than adults, with at least 2/3 suffering long term sequels such as developmental (motor, global intellectual, language...) and behavioral disabilities, epilepsy, and low adaptative and academic skills...

Stenotic cerebral arteriopathy is identified as AIS etiology in 60-80% of previously healthy children and the course of this arteriopathy is the strongest predictor of recurrent events. 30-40% of these children have a focal unilateral cerebral arteriopathy (FCA). Childhood FCA is suspected to be an inflammatory vessel wall pathology triggered by varicella and other (viral) infections. As recurrences occur for the great majority in the first 6 months after the index event, aspirin 5 mg/kg/day is recommended for at least 18 months to 2 years.

As there is a rational for using immunomodulatory drugs at the acute stage of FCA, immunotherapies are currently used by neuropaediatricians in AIS, mainly as steroids for children with stenosing arteriopathies. However, due to weak evidences, the literature cannot either encourage or discourage this practice.

The long term course of children with FCA is only approach to date by retrospective studies and controversies about outcome remain (for example, the recurrence risk on antithrombotic treatment varies notably from quasi zero to 25%). And finally, it is shown in childhood stroke, as well as in the global field of longstanding impairment, that parental and medical points of view do not match consistently. Longitudinal studies are needed to deserve this familial approach.

ELIGIBILITY:
Inclusion Criteria:

-- Aged 6 months to <15 years

* AIS ≤ 48 hours

  * Newly acquired focal neurological deficit with confirmation by magnetic resonance imaging (MRI) of ischaemic lesion in an arterial territory corresponding with the clinical features (definition of Arterial ischemic stroke).
  * Magnetic resonance arteriography showing unilateral proximal stenosis or irregularities of the corresponding carotid trifurcation (i.e. terminal carotid and/or M1-M2 and/or A1 segments) or of the posterior circulation (P1-P2 segments).
  * No evidence of an underlying systemic disorder (e.g. lupus erythematodes) explaining the features.
  * Informed and signed consent of parents or legal guardians.
* French Social Security (Sécurité sociale; i.e. national health coverage) affiliation

Exclusion Criteria:

* Children with secondary central nervous system angiitis due to infections (meningitis, endocarditis, borreliosis), rheumatic or other systemic inflammatory diseases (e.g. lupus erythematodes). These children are already under immune suppression or need other co-medications regarding their underlying disease.
* Children with known syndromal and/or genetic vasculopathies such as phaces syndrome, Neurofibromatosis type 1, trisomy 21.
* Children with moyamoya or sickle cell disease.
* Children with a progressive large to medium vessel childhood primary angiitis of the central nervous system with two out of the following three criteria : Children with progressive neurocognitive dysfunction; Children with bilateral lesions/vessel involvement; Children with distal arterial stenosis (beyond the M2, A1 or P2 segment).

  - Children already on steroid treatment at disease onset or with a contraindication to receive steroid treatment (e.g. congenital or acquired immunodeficiency).
* Children with delayed diagnosis ≥3 days as treatment start is not allowed to be more ≥5 day-delayed.
* Contraindications to steroids (see also summary of product characteristics in chapter 1.1) and notably: Not-manageable infectious, hydro-electrolytic or metabolic (e.g. diabetes mellitus) disorders, or elevated blood pressure, Serious behavioral disorders, Current vaccination with live or attenuated live strains, Allergy/sensibility to any ingredient, Association with some medications such as antiarrhythmic drugs.

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to recovery up to 12 months | Up to 12 months
  Evaluate of time to recovery up to 12 months by score paediatric Recurrence and Recovery Questionnaire (RRQ )

SECONDARY OUTCOMES:
Improvement of functional outcome by face-to-face visits | Months:1,6,12, 24 and 36
  Evaluate of Improvement of functional outcome by face-to-face visits by score Paediatric Stroke Outcome Measure (PSOM), modified Rankin Scale (mRS) and Vineland Adaptive Behaviour Scale (VABS).
Arteriopathic course along time | Months: 1, 6, 24
  Evaluate of Arteriopathic course along time by comparison between magnetic resonance (MR) arteriography and initial imaging.
Recurrence of stroke, epilepsy, neurological and developmental sequels, and academic achievement | Months: 1, 3, 6,12, 24 and 36
  Evaluate recurrence of stroke, epilepsy, neurological and developmental sequels, and academic achievement at 6, 12, 24 and 36 months. Neurological outcome will be assessed by standard clinical examination: motricity, sensibility, coordination, oculomotricity and visual field, cranial nerves…
Outcome by age group | Months 72
  Evaluate outcome by age group. All endpoints will be stratified for the whole cohort by the following age group: 0.5-3 years; 3-6 years; 6-10 years and ≥10 years. This will be done in a centrally-manner at Clinical Trials Unit (CTU) Bern.
Familial impact | Months 72
  Evaluate of familial impact by Alberta Perinatal Stroke Parental Outcome Measure (APSOM) and indepth interview through semi-structured interviews. The objective is to report the lived experience of parents whose child was included in the study.
Number of serious adverse events | Months 72
  Analysis of number of serious adverse events and their cause, consequence.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane CHABRIER, MD, Principal Investigator — CHU SAINT-ETIENNE

IPD SHARING:
Plan to Share IPD: No